CLINICAL TRIAL: NCT01276379
Title: Single-Arm, Multicenter, Prospective, Phase 2 Study for the Evaluation of Biomarkers in Patients With Advanced &/or Metastatic Colorectal Cancer With Wild Type KRAS Treated Biweekly With Chemotherapy and Cetuximab as First-Line Treatment
Brief Title: Study Evaluating Biomarkers in Patients With Colorectal Cancer and Native KRAS Treated With Chemotherapy + Cetuximab
Acronym: POSIBA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Grupo Espanol Multidisciplinario del Cancer Digestivo (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: GEMCAD-1002; 2010-019236-12 (EudraCT Number)
Record Dates: First submitted 2011-01-12; First posted 2011-01-13 (Estimated); Results first posted 2021-07-02 (Actual); Last update posted 2021-07-02 (Actual); Status verified 2021-06

CONDITIONS: Colorectal Cancer
Keywords: colorectal cancer; advanced; metastatic; KRAS; biomarkers (BRAF, IGF1P/MMp7,PI3K-PTEN); cetuximab
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis; Hereditary Sensory and Autonomic Neuropathies | interventions — Leucovorin; Fluorouracil; Irinotecan; Oxaliplatin; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- FOLFIRI (m) or FOLFOX-6 (m) + cetuximab (Experimental): FOLFOX/FOLFIRI + cetuximab 500mg/m2 bi-weekly for 6 months, then bi-weekly cetuximab as monotherapy.
  Interventions: Drug: FOLFIRI (m); Drug: FOLFOX-6 (m); Drug: Cetuximab

INTERVENTIONS:
Drug: FOLFIRI (m) — FOLFIRI (m) chemotherapy will be administered on day 1 of each 14-days-cycle. The administered doses will be:
  * Irinotecan 180 mg/m2 in infusion i.v., 120 minutes, on day 1 of each cycle.
  * l-Leucovorin 200 mg/m2 (or d,l-leucovorin 400 mg/m2), in infusion i.v., 120 minutes, on day 1.
  * One bolus i.v. (2-4 minutes) of 400 mg/m2 of 5-FU on day 1.
  * 5-FU in continuous infusion (2400 mg/m2) administered through an ambulatory pump during 46-48 hours.
  Other Names: folinic acid, fluorouracil and irinotecan.
Drug: FOLFOX-6 (m) — FOLFOX6 (m) chemotherapy will be administered on day 1 of each 14-days-cycle. The administered doses will be:
  * Oxaliplatin 85 mg/m2 in infusion i.v., 120 minutes, on day 1 of each cycle.
  * l-Leucovorin 200 mg/m2 (or d,l-leucovorin 400 mg/m2) in infusion i.v., 120 minutes, on day 1.
  * One bolus i.v. (2-4 minutes) of 400 mg/m2 of 5-FU on day 1.
  * 5-FU in continuous infusion (2400 mg/m2) administered through an ambulatory pump during 46-48 hours.
  Other Names: folinic acid, fluorouracil and oxaliplatin.
Drug: Cetuximab — - 500 mg/m2 i.v. Every 2 weeks.
  Other Names: erbitux

SUMMARY:
Advanced colorectal cancer (ACRC) is a heterogeneous disease and classification of patients is nowadays inefficient. Roughly twenty per cent of patients present with favorable figures (less than 4 liver nodules and less than 5 cm) and are suitable for local treatments (surgery or local-ablative therapies). Additionally, 10-15% of patients have poor performance status (PS >2) or are severe disabled due to geriatric syndromes or/and co-morbid diseases that preclude any treatment strategies than best supportive care alone. The rest of patients (fit patients not suitable for radical treatments) constitute the population of patients treated with palliative therapies. Despite of it not all these patients have the same prognosis. Patients with PS 0,1 and levels of LDH <ULN (Intermediate-risk patients) have better PFS and OS irrespective of therapy in all randomized clinical trials (de Gramont et al, JCO 2000; Douillard et al, Lancet 2000; Koopman et al, 2007).

CRYSTAL trial shows a benefit in PFS (1.5 months) in RASWT of FOLFIRI plus cetuximab compared with FOLFIRI alone. Nowadays the selection of patients for cetuximab treatment is based on mutational status of KRAS, which allow to select those patients who will not respond to therapy. Other surrogate markers of activity should be also evaluated. Our hypothesis is that the suggested biomarkers will allow the selection of the patients who will benefit the most from the biweekly cetuximab treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age ≥ 18 years
* Able to sign an informed consent form
* Advanced and/or metastatic colorectal cancer
* Colorectal cancer with KRAS wild type genotype
* At least one unidimensionally measurable lesion according to RECIST criteria (1.1 revised) (to be assessed ≤ 28 days prior to the study treatment)
* All patients with the following features will be included:

  1. Progression free survival > 6 months after adjuvant treatment +/- radiotherapy
  2. "De novo" diagnosis of the disease
* Performance ECOG status of 0-2
* Life expectancy ≥ 3 months
* Adequate bone marrow function: neutrophils ≥1,5 x 10^9/L; platelets ≥ 100 x 10^9/L; hemoglobin ≥9 g/dL.
* Adequate liver, renal and hematological function as follows:

  1. Adequate liver function: SGOT and SGPT 2.5 x ULN (5 x ULN in case of hepatic metastasis). Total bilirubin < 1,5 x ULN. Alkaline phosphatase 2,5 x LSN (5 x ULN if hepatic metastasis or 10 x ULN if bone metastasis)
  2. Creatinine clearance or creatinine clearance during 24 hours ≥ 50 mL/min
  3. Magnesium ≥ LLN, calcium ≥ LLN

Exclusion Criteria:

* PS > 2 or elderly patients with fragility criteria
* Previous surgery for metastasis
* Previous systemic treatment for the metastatic colorectal cancer
* Previous treatment with antibodies anti-EGFR or treatment with small-molecule EGFR tyrosine kinase inhibitors or EGFR signal transduction inhibitors. Subjects who suspend their first dose due to a reaction to the infusion can participate
* Central nervous system metastasis (except: treated subjects with asymptomatic CNS metastasis who have not received steroids within the 30 days prior to inclusion)
* Prior malignant tumor in the last 5 years, except: basal cell carcinoma of the skin or pre-invasive cervical cancer
* Unresolved toxicities from a prior systemic treatment which do not qualify the patient for inclusion
* Presence of peripheral neuropathy (degree > 1 in the ctc version 3.0) and serious nonhealing wound, ulcer, or bone fracture
* Hormonal treatment, immunotherapy or experimental or approved antibodies/proteins ≤ 30 days before the inclusion
* Uncontrolled serious cardiovascular disease or: congestive cardiac failure NYHA lll or lV, unstable angina pectoris, myocardial infarction precedents in the past 12 months, significant arrhythmias
* Interstitial pneumonitis or pulmonary fibrosis precedents, or interstitial pneumonitis or pulmonary fibrosis signs on the thoracic CT-scan
* Treatment for systemic infection within the 14 days prior to treatment
* Acute/subacute intestinal occlusion and/or active inflammatory bowel disease or any other bowel disease producing chronic diarrhea
* Precedent of Gilbert's syndrome or dihydropyrimidine dehydrogenase deficiency
* Precedent of any disease which can increase the risks associated to the participation in the study or interfere in the study results
* Known positive test for the following infections: HIV, Hepatitis C + abnormal liver enzymes values, active chronic Hepatitis B (except Hepatitis C seropositive with normal liver enzymes)
* All concurrent diseases which can increase the toxicity risk
* The individual presents a disorder of any kind which jeopardizes their ability to give their written consent form and/or fulfill the study procedures
* Any investigational agent within 30 days before enrolment
* Pregnant or breastfeeding woman, or planning to get pregnant within the 6 months after treatment
* Surgery (excluding the diagnostic biopsy or placing of a central venous catheter)
* Woman or man of childbearing potential not consenting to use adequate contraceptive precautions during the study and 6 months after de last administration for women, and 1 month for men
* Unability to fulfill the study requirements by the patients
* Psychological, family, sociological or geographical conditions that may interfere with the fulfillment of the study protocol and the follow-up calendar

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 221 (Actual)
Dates: Start 2011-01; Primary Completion 2017-03-15 (Actual); Study Completion 2017-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jesús García Foncillas, MD, Study Chair — Grupo Espanol Multidisciplinario del Cancer Digestivo; Xavier García-Albeniz, MD, Study Chair — Grupo Espanol Multidisciplinario del Cancer Digestivo
Locations (27):
- Spain (27):
  - Hospital Provincial de Castellón, Castellon, Castellón
  - Hospital Son Espases, Palma, Malllorca
  - Hospital Son Llàtzer, Palma, Mallorca
  - Hospital Sant Joan de Reus, Reus, Tarragona
  - Complejo Hospitalario Universitario de Albacete, Albacete
  - Hospital Infanta Cristina de Badajoz, Badajoz
  - Hospital de Barbastro, Barbastro
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital General Yagüe, Burgos
  - Hospital Sant Jaume de Calella, Calella
  - Hospital San Pedro de Alcántara, Cáceres
  - Hospital General Universitario de Elche, Elche
  - Hospital de Jaén, Jaén
  - Hospital Universitario de Gran Canaria Dr. Negrín, Las Palmas de Gran Canaria
  - Hospital Universitari Arnau de Vilanova de Lleida, Lleida
  - Fundación Jimenez Díaz, Madrid
  - Hospital de Móstoles, Madrid
  - Hospital Universitario la Paz, Madrid
  - Hospital de Mataró, Mataró
  - Clínica Universitaria de Navarra, Pamplona
  - Hospital de Navarra, Pamplona
  - Hospital de Sagunto, Sagunto
  - Mutua de Terrassa, Terrassa
  - Hospital Virgen de la Salud, Toledo
  - Instituto Valenciano de Oncología, Valencia
  - Hospital Clínico Universitario Lozano Blesa, Zaragoza
  - Hospital Miguel Servet, Zaragoza

REFERENCES:
- [Derived] Maurel J, Alonso V, Escudero P, Fernandez-Martos C, Salud A, Mendez M, Gallego J, Rodriguez JR, Martin-Richard M, Fernandez-Plana J, Manzano H, Mendez JC, Zanui M, Falco E, Gil-Raga M, Aparicio J, Feliu J, Garcia-Albeniz X, Torres F, Rojo F, Bellosillo B, Mendiola M, Fernandez V, Reig O, Claes B, Maertens G, Sablon E, Jacobs B, Montagut C. Clinical Impact of Circulating Tumor RAS and BRAF Mutation Dynamics in Patients With Metastatic Colorectal Cancer Treated With First-Line Chemotherapy Plus Anti-Epidermal Growth Factor Receptor Therapy. JCO Precis Oncol. 2019 Dec;3:1-16. doi: 10.1200/PO.18.00289. PMID 35100697
- [Derived] Garcia-Albeniz X, Alonso V, Escudero P, Mendez M, Gallego J, Rodriguez JR, Salud A, Fernandez-Plana J, Manzano H, Zanui M, Falco E, Feliu J, Gil M, Fernandez-Martos C, Bohn U, Alonso C, Calderero V, Rojo F, Cuatrecasas M, Maurel J. Prospective Biomarker Study in Advanced RAS Wild-Type Colorectal Cancer: POSIBA Trial (GEMCAD 10-02). Oncologist. 2019 Nov;24(11):e1115-e1122. doi: 10.1634/theoncologist.2018-0728. Epub 2019 Jun 24. PMID 31235483
- See also: GEMCAD group — http://www.gemcad.es/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All patients were allocated in the same treatment arm. Some patient characteristics and results may be reported according to the mutational status of the patients despite all patients received the same treatment schedule
Groups:
- FOLFIRI (m) or FOLFOX-6 (m) + Cetuximab: FOLFOX/FOLFIRI + cetuximab 500mg/m2 bi-weekly for 6 months, then bi-weekly cetuximab as monotherapy.
  FOLFIRI (m): FOLFIRI (m) chemotherapy will be administered on day 1 of each 14-days-cycle. The administered doses will be:
  * Irinotecan 180 mg/m2 in infusion i.v., 120 minutes, on day 1 of each cycle.
  * l-Leucovorin 200 mg/m2 (or d,l-leucovorin 400 mg/m2), in infusion i.v., 120 minutes, on day 1.
  * One bolus i.v. (2-4 minutes) of 400 mg/m2 of 5-FU on day 1.
  * 5-FU in continuous infusion (2400 mg/m2) administered through an ambulatory pump during 46-48 hours.
  FOLFOX-6 (m): FOLFOX6 (m) chemotherapy will be administered on day 1 of each 14-days-cycle. The administered doses will be:
  * Oxaliplatin 85 mg/m2 in infusion i.v., 120 minutes, on day 1 of each cycle.
  * l-Leucovorin 200 mg/m2 (or d,l-leucovorin 400 mg/m2) in infusion i.v., 120 minutes, on day 1.
  * One bolus i.v. (2-4 minutes) of 400 mg/m2 of 5-FU on day 1.
  * 5-FU in continuous infusion (2400 mg/m2) administered through an ambulatory pump during 46-48 hours.
  Cetuximab: - 500 mg/m2 i.v. Every 2 weeks.
Period: Overall Study
Arm/Group | FOLFIRI (m) or FOLFOX-6 (m) + Cetuximab
Started | 221
Completed | 181
Not Completed | 40
Not completed — Screening failure | 40

BASELINE CHARACTERISTICS:
Population: Evaluable patients
Groups:
- WT BRAF - FOLFIRI (m) or FOLFOX-6 (m) + Cetuximab: Patients with a determination of BRAF status and presence of Wild type (WT) BRAF gen.
  FOLFOX/FOLFIRI + cetuximab 500mg/m2 bi-weekly for 6 months, then bi-weekly cetuximab as monotherapy.
  FOLFIRI (m): FOLFIRI (m) chemotherapy will be administered on day 1 of each 14-days-cycle. The administered doses will be:
  * Irinotecan 180 mg/m2 in infusion i.v., 120 minutes, on day 1 of each cycle.
  * l-Leucovorin 200 mg/m2 (or d,l-leucovorin 400 mg/m2), in infusion i.v., 120 minutes, on day 1.
  * One bolus i.v. (2-4 minutes) of 400 mg/m2 of 5-FU on day 1.
  * 5-FU in continuous infusion (2400 mg/m2) administered through an ambulatory pump during 46-48 hours.
  FOLFOX-6 (m): FOLFOX6 (m) chemotherapy will be administered on day 1 of each 14-days-cycle. The administered doses will be:
  * Oxaliplatin 85 mg/m2 in infusion i.v., 120 minutes, on day 1 of each cycle.
  * l-Leucovorin 200 mg/m2 (or d,l-leucovorin 400 mg/m2) in infusion i.v., 120 minutes, on day 1.
  * One bolus i.v. (2-4 minutes) of 400 mg/m2 of 5-FU on day 1.
  * 5-FU in continuous infusion (2400 mg/m2) administered through an ambulatory pump during 46-48 hours.
  Cetuximab: - 500 mg/m2 i.v. Every 2 weeks.
- Mutant BRAF - FOLFIRI (m) or FOLFOX-6 (m) + Cetuximab: Patients with a determination of BRAF status and presence of a mutation in the BRAF gen.
  FOLFOX/FOLFIRI + cetuximab 500mg/m2 bi-weekly for 6 months, then bi-weekly cetuximab as monotherapy.
  FOLFIRI (m): FOLFIRI (m) chemotherapy will be administered on day 1 of each 14-days-cycle. The administered doses will be:
  * Irinotecan 180 mg/m2 in infusion i.v., 120 minutes, on day 1 of each cycle.
  * l-Leucovorin 200 mg/m2 (or d,l-leucovorin 400 mg/m2), in infusion i.v., 120 minutes, on day 1.
  * One bolus i.v. (2-4 minutes) of 400 mg/m2 of 5-FU on day 1.
  * 5-FU in continuous infusion (2400 mg/m2) administered through an ambulatory pump during 46-48 hours.
  FOLFOX-6 (m): FOLFOX6 (m) chemotherapy will be administered on day 1 of each 14-days-cycle. The administered doses will be:
  * Oxaliplatin 85 mg/m2 in infusion i.v., 120 minutes, on day 1 of each cycle.
  * l-Leucovorin 200 mg/m2 (or d,l-leucovorin 400 mg/m2) in infusion i.v., 120 minutes, on day 1.
  * One bolus i.v. (2-4 minutes) of 400 mg/m2 of 5-FU on day 1.
  * 5-FU in continuous infusion (2400 mg/m2) administered through an ambulatory pump during 46-48 hours.
  Cetuximab: - 500 mg/m2 i.v. Every 2 weeks.
- Total: Total of all reporting groups
Arm/Group | WT BRAF - FOLFIRI (m) or FOLFOX-6 (m) + Cetuximab | Mutant BRAF - FOLFIRI (m) or FOLFOX-6 (m) + Cetuximab | Total
Number analyzed (Participants) | 161 | 20 | 181
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62 (10.5) | 67 (7.4) | 65 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 7 | 53
  Male | 115 | 13 | 128
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 161 | 20 | 181
Region of Enrollment [Number; unit: participants]
  Spain | 161 | 20 | 181
Stage [Count of Participants; unit: Participants] — The stage of a cancer describes the size and spread of a tumour:
  stage I - The cancer has grown through the mucosa and has invaded the muscular layer of the colon or rectum.
  stage II - The cancer has grown through the wall of the colon or rectum stage III - The cancer has grown through the inner lining or into the muscle layers of the intestine. It has spread to lymph nodes stage IV - The cancer has spread to a distant part of the body
  Participants
    Stage I | 1 | 0 | 1
    Stage II | 13 | 0 | 13
    Stage III | 30 | 5 | 35
    Stage IV | 117 | 15 | 132
Primary location [Count of Participants; unit: Participants] — Part of the colon where the primary tumor was located
  Participants
    Ascending colon | 23 | 9 | 32
    Transverse colon | 12 | 2 | 14
    Descending colon | 10 | 4 | 14
    Sigmoid colon | 73 | 3 | 76
    Rectum | 43 | 2 | 45
Surgery of the primary tumor [Count of Participants; unit: Participants] — Percentage of patients that had surgery for their primary colorectal tumor
  Participants | 91 | 10 | 101
Performance Status (PS) [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group (ECOG) performance status. ECOG scale measures the performance status of a patients. It ranges from 0 (fully active, able to carry on all pre-disease performance without restriction) to 5 (death).
  Participants
    ECOG 0 | 112 | 7 | 119
    ECOG 1 | 49 | 13 | 62
Number of metastatic organs [Count of Participants; unit: Participants] — Percentage of patients presenting metastasis in one or more distant organs. The number of patients with 1,2, 3 or more than 4 affected organs are reported
  Participants
    1 | 87 | 7 | 94
    2 | 58 | 11 | 69
    3 | 15 | 2 | 17
    4 or higher | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: Measurements according to RECIST 1.1 criteria (Response Evaluation Criteria in Solid Tumors). Main techniques: CT-scan. Two groups will be defined based on the score built from the proposed clinical variables and biomarkers. Instead of a binomial distribution, a Log-rank method has been used to calculate the sample size in order to include all the incidents during the follow-up. Expecting a minimum 20% difference (60 vs. 40%) on PFS at 12 months between groups and with the following assumptions:
  Alpha error (bilateral): 5% Beta error: 20% Results are reported by subgroups to compare outcome measure according to BRAF mutation. All patients belong to same treatment/study arm.
Time Frame: 4 years
Population: Evaluable population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | WT BRAF - FOLFIRI (m) or FOLFOX-6 (m) + Cetuximab | Mutant BRAF - FOLFIRI (m) or FOLFOX-6 (m) + Cetuximab
Number analyzed (Participants) | 161 | 20
Months | 11.4 [9.9 to 13.1] | 5.9 [3.3 to 7.8]
Statistical Analysis 1: Comparison: WT BRAF - FOLFIRI (m) or FOLFOX-6 (m) + Cetuximab vs Mutant BRAF - FOLFIRI (m) or FOLFOX-6 (m) + Cetuximab; Test type: Superiority; p = 0.004, Log Rank; Hazard Ratio (HR) = 2.01, 95% CI 2-sided [1.23 to 3.29]

2. Secondary Outcome: Overall Survival
Description: Measured as time in months from start of study treatment to death or lost to follow up.
  Results are reported by subgroups to compare outcome measure according to BRAF mutation. All patients belong to same treatment/study arm.
Time Frame: 4 years
Population: Evaluable population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | WT BRAF - FOLFIRI (m) or FOLFOX-6 (m) + Cetuximab | Mutant BRAF - FOLFIRI (m) or FOLFOX-6 (m) + Cetuximab
Number analyzed (Participants) | 161 | 20
Months | 32.6 [27.5 to 38.8] | 9.3 [5.3 to 22]
Statistical Analysis 1: Comparison: WT BRAF - FOLFIRI (m) or FOLFOX-6 (m) + Cetuximab vs Mutant BRAF - FOLFIRI (m) or FOLFOX-6 (m) + Cetuximab; Test type: Superiority; p < 0.0001, Log Rank; Hazard Ratio (HR) = 2.29, 95% CI 2-sided [1.33 to 3.96]

3. Secondary Outcome: Response Duration
Description: Duration of the partial or total response to the treatment. Evaluation and classification according to RECIST 1.1 criteria (Response Evaluation Criteria in Solid Tumors)
Time Frame: 4 years
Population: Evaluable population
Measure: Median (Full Range); unit: Months
Arm/Group | FOLFIRI (m) or FOLFOX-6 (m) + Cetuximab
Number analyzed (Participants) | 181
Months | 8.66 [1.16 to 53.49]

4. Secondary Outcome: Frequency of Adverse Events
Description: Frequency and type of adverse events (AEs). AEs were coded according to NCI CTCAE V3.0 and classified by frequency, relatedness to study treatment (related/not related) and severity (Grade).
  Severity ranges from grade 1 (low intensity) to Grade 5 (max. intensity, death)
Time Frame: 4 years
Population: Safety population (all patients that received at least one infusion of study treatment)
Measure: Count of Participants; unit: Participants
Arm/Group | FOLFIRI (m) or FOLFOX-6 (m) + Cetuximab
Number analyzed (Participants) | 218
Participants
  Any AEs: yes | 198
  Any AEs: no | 20
  Grade 3 or higher AEs: yes | 138
  Grade 3 or higher AEs: no | 80
  Grade 5 AEs: yes | 5
  Grade 5 AEs: no | 213
  Treatment related AEs of any grade: yes | 176
  Treatment related AEs of any grade: no | 42
  Treatment related AEs grade 3 or higher: yes | 101
  Treatment related AEs grade 3 or higher: no | 117

5. Secondary Outcome: Secondary Biomarkers Analysis
Description: The secondary biomarkers in serum and tumoral tissue will be analysed in order to predict the acquired resistance.
Time Frame: 4 years
Population: Evaluable population
Measure: Count of Participants; unit: Participants
Arm/Group | FOLFIRI (m) or FOLFOX-6 (m) + Cetuximab
Number analyzed (Participants) | 181
Participants
  PI3K and PTEN: WT | 69
  PI3K and PTEN: Mutant | 98
  PI3K and PTEN: UK | 14
  IGF-1RP/MMP7: WT | 158
  IGF-1RP/MMP7: Mutant | 23
  IGF-1RP/MMP7: UK | 0

6. Secondary Outcome: Tumoral Response
Description: Measurements according to RECIST 1.1 criteria (Response Evaluation Criteria in Solid Tumors). Main techniques: CT-scan. Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR Results are reported by subgroups to compare outcome measure according to BRAF mutation. All patients belong to same treatment/study arm.
Time Frame: 4 years
Population: Evaluable population
Measure: Count of Participants; unit: Participants
Arm/Group | WT BRAF - FOLFIRI (m) or FOLFOX-6 (m) + Cetuximab | Mutant BRAF - FOLFIRI (m) or FOLFOX-6 (m) + Cetuximab
Number analyzed (Participants) | 161 | 20
Participants
  Complete response (CR) | 16 | 1
  Partial response (PR) | 106 | 6
  Stable disease (SD) | 25 | 6
  Progression disease (PD) | 8 | 4
  Not evaluable (NE) | 6 | 3

ADVERSE EVENTS:
Time Frame: 4 years
Description: Safety assessments included patient history and physical examinations, vital signs, ECOG PS, AEs, blood chemistry, and blood counts, which were performed at each visit.
  AE severity was graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), version 3.0. Relation to cetuximab or chemotherapy (definitely, probably, possibly, unlikely, or unrelated) were assessed by the PI.
  AEs reported by treatment arm, which includes all patients
Arm/Group | FOLFIRI (m) or FOLFOX-6 (m) + Cetuximab
All-Cause Mortality (participants affected / at risk) | 136/218
Serious Adverse Events (participants affected / at risk) | 173/218
Other Adverse Events (participants affected / at risk) | 198/218
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FOLFIRI (m) or FOLFOX-6 (m) + Cetuximab (N=218)
Alopecia (Skin and subcutaneous tissue disorders) | 4 (4)
Anemia (Blood and lymphatic system disorders) | 4 (4)
Anorexia (Metabolism and nutrition disorders) | 2 (2)
Ascites (Gastrointestinal disorders) | 1 (1)
Asthenia (General disorders) | 19 (19)
Diarrhoea (Gastrointestinal disorders) | 28 (28)
Pain (General disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
Edema (General disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Fever (General disorders) | 1 (1)
Fistula (Gastrointestinal disorders) | 7 (7)
Hepatic toxicity (Hepatobiliary disorders) | 3 (3)
Infections (Infections and infestations) | 9 (9)
Leucocytopenia (Blood and lymphatic system disorders) | 4 (4)
Mucositis (Gastrointestinal disorders) | 14 (14)
Nausea (Gastrointestinal disorders) | 9 (9)
Neuropathy (Nervous system disorders) | 5 (5)
Neutropenia (Blood and lymphatic system disorders) | 53 (53)
Febrile neutropenia (Blood and lymphatic system disorders) | 5 (5)
Intestinal obstruction (Gastrointestinal disorders) | 10 (10)
Ocular alterations non otherwise specified (NOS) (Eye disorders) | 1 (1)
paresthesia (Nervous system disorders) | 5 (5)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3)
Alergic reaction (Immune system disorders) | 7 (7)
Skin reaction (Skin and subcutaneous tissue disorders) | 29 (29)
rectal bleeding (Gastrointestinal disorders) | 1 (1)
Hand-foot syndrome (General disorders) | 1 (1)
Transaminitis (Hepatobiliary disorders) | 2 (2)
Cardiac disorders NOS (Cardiac disorders) | 2 (2)
Metabolic disorders NOS (Metabolism and nutrition disorders) | 6 (6)
Gastrointestinal disorders NOS (Gastrointestinal disorders) | 5 (5)
General and site reactions NOS (General disorders) | 2 (2)
Muscolosqueletal disorders NOS (Musculoskeletal and connective tissue disorders) | 5 (5)
Ocular disorders NOS (Eye disorders) | 3 (3)
Urinary disorders NOS (Renal and urinary disorders) | 4 (4)
Respiratory disorders NOS (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Vascular disorders NOS (Vascular disorders) | 10 (10)
Xerosis (Skin and subcutaneous tissue disorders) | 8 (8)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FOLFIRI (m) or FOLFOX-6 (m) + Cetuximab (N=218)
Alopecia (Skin and subcutaneous tissue disorders) | 29 (29)
Anemia (Blood and lymphatic system disorders) | 34 (34)
Anorexia (Metabolism and nutrition disorders) | 27 (27)
Asthenia (General disorders) | 101 (101)
Diarrhoea (Gastrointestinal disorders) | 80 (80)
Dysgeusia (Nervous system disorders) | 22 (22)
Pain NOS (General disorders) | 21 (21)
Abdominal pain (Gastrointestinal disorders) | 28 (28)
Constipation (Gastrointestinal disorders) | 40 (40)
Fever (General disorders) | 25 (25)
Fistula (Gastrointestinal disorders) | 47 (47)
Infections NOS (Infections and infestations) | 17 (17)
Leucopenia (Blood and lymphatic system disorders) | 16 (16)
Mucositis (Gastrointestinal disorders) | 87 (87)
Nausea (Gastrointestinal disorders) | 60 (60)
Neuropathy (Nervous system disorders) | 72 (72)
Neutropenia (Blood and lymphatic system disorders) | 37 (37)
Paresthesia (Nervous system disorders) | 45 (45)
Thrombocytopenia (Blood and lymphatic system disorders) | 22 (22)
Cutaneous reaction (Skin and subcutaneous tissue disorders) | 134 (134)
Mucosa dryness (Gastrointestinal disorders) | 13 (13)
Transaminitis (Hepatobiliary disorders) | 13 (13)
Metabolic disorders NOS (Metabolism and nutrition disorders) | 36 (36)
gastrointestinal disorders (Gastrointestinal disorders) | 40 (40)
Musculoskeletal disorders NOS (Musculoskeletal and connective tissue disorders) | 20 (20)
Ocular disorders NOS (Eye disorders) | 24 (24)
Psychiatric disorders NOS (Psychiatric disorders) | 12 (12)
Urinary disorders NOS (Renal and urinary disorders) | 13 (13)
Respiratory disorders NOS (Respiratory, thoracic and mediastinal disorders) | 29 (29)
Vascular disorders NOS (Vascular disorders) | 12 (12)
trichomegaly (Congenital, familial and genetic disorders) | 11 (11)
Xerosis (Skin and subcutaneous tissue disorders) | 36 (36)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Complying with the R.D. 223/2004, the results of this trial will be published, both positive and negative results in recognized scientific journals or congress.

The Sponsor and the Investigators are fully committed to publishing the results of the study.

All publications (i.e., manuscripts, abstracts, oral / slide presentations, book chapters) based on this study must be submitted to the sponsor for review prior to publication.

DOCUMENTS (2):
  • Study Protocol (2010-02-23): https://cdn.clinicaltrials.gov/large-docs/79/NCT01276379/Prot_000.pdf
  • Statistical Analysis Plan (2011-06-27): https://cdn.clinicaltrials.gov/large-docs/79/NCT01276379/SAP_001.pdf